CLINICAL TRIAL: NCT01235897
Title: A Phase Ib Dose-escalation Trial of the AKT Inhibitor MK2206 in Combination With Weekly Paclitaxel With or Without Trastuzumab
Brief Title: MK-2206, Paclitaxel and Trastuzumab in Treating Patients With HER2-overexpressing Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10998
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Advanced Solid Tumors; Tumors; Cancer
Keywords: Neoplasms; Paclitaxel; Trastuzumab
MeSH Terms: conditions — Neoplasms | interventions — MK 2206; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maximum tolerated dose (Experimental)
  Interventions: Drug: MK-2206; Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: MK-2206 — Different dose levels of MK-2206 will studied, and co-administered with paclitaxel and trastuzumab. MK-2206 will be given orally with a starting dose of 135 mg weekly
Drug: Paclitaxel — 80 mg/m2 weekly - paclitaxel
Drug: Trastuzumab — 2 mg/kg weekly after a 1-time loading dose of 4 mg/kg - trastuzumab
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to test the safety and safest highest dose of an investigational drug called MK-2206 when given in combination with paclitaxel and trastuzumab in patients with Human Epidermal growth factor Receptor 2 (HER2)-overexpressing solid tumor malignancies.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and maximum tolerated dose (MTD) of MK-2206 in combination with paclitaxel and trastuzumab when given to patients with HER2-overexpressing solid tumor malignancies. MK-2206 is an oral drug (taken by mouth) that turns off a protein called AKT inside cancer cells. This could be helpful in treating treatment-resistant cancers, because AKT allows cells to survive despite active anticancer treatment. In the case of HER2-positive cancers, laboratory studies suggest that the drug combination of MK-2206 and paclitaxel and trastuzumab may be effective.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-confirmed metastatic or locally advanced, unresectable HER2+ cancer. HER2+ will be defined as 3+ expression by immunohistochemistry (IHC) OR >2-fold gene amplification by Fluorescence In Situ Hybridization (FISH).
2. Male or female and ≥18 years of age on the day of signing informed consent.
3. Performance status of 0-2 on the ECOG Performance Scale and life expectancy > 3 months.
4. Have evaluable disease. Measureable disease is not required
5. Adequate organ function as indicated by the following laboratory values:

   * Absolute neutrophil count (ANC) = ≥1,500 /μL
   * Platelets = ≥100,000 /μL
   * Hemoglobin = ≥9 g/dL
   * Serum creatinine = ≤1.5 x upper limit of normal (ULN) OR calculated creatinine clearance = ≥60 mL/min for patients with creatinine levels >1.5 x institutional ULN
   * Serum total bilirubin = ≤1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 x ULN
   * AST (SGOT) and ALT (SGPT) = ≤2.5 x ULN
   * Prothrombin time (PT)/INR = ≤1.2 x ULN
   * Partial thromboplastin time (PTT) = ≤1.2 x ULN
   * Fasting serum glucose = ≤126 mg/dl
   * Hemoglobin A1c (HgbA1c) = ≤7%
   * Potassium = in normal range
6. Female patient of childbearing potential must test negative for pregnancy and agree to the use of effective methods of contraception while on study.
7. Voluntarily agree to participate by giving written informed consent.
8. Able to swallow capsules and has no surgical or anatomical condition that will prevent the patient from swallowing and absorbing oral medications on an ongoing basis.
9. Prior taxane, trastuzumab, lapatinib, and other HER2 directed therapy in the adjuvant or metastatic setting is allowed.
10. Any number of prior lines of chemotherapy in the metastatic setting is allowed.
11. Concomitant use of bisphosphonates is allowed.
12. Patients with stable and clinically insignificant central nervous system (CNS) disease are allowed. Patients must be off steroids with no new CNS symptoms or findings on radiographic imaging for 1 month.

Exclusion Criteria:

1. Patient who has had chemotherapy, radiotherapy, or hormonal therapy within 3 weeks (6 weeks for nitrosoureas, mitomycin C or bevacizumab), or who has not recovered from the adverse events due to previous agents administered more than 4 weeks prior to Study Day 1. Patient must not have received trastuzumab or lapatinib within 2 weeks of study Day 1. If the patient has residual toxicity from prior treatment, toxicity must be ≤ Grade 1.
2. Less than 4 weeks post major surgical procedure (defined as one that required general anesthesia)(all surgical wounds must be fully healed).
3. Currently participating or has participated in a study with an investigational compound or device within 30 days of Study Day 1.
4. Known active CNS metastases and/or carcinomatous meningitis. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 1 month prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis (2) off steroids that are used to minimize surrounding brain edema. Patients with clinically insignificant brain metastases that do not require treatment are eligible.
5. Has a primary central nervous system tumor.
6. Known hypersensitivity to the components of study drug or its analogs.
7. History or current evidence of clinically significant heart disease including:

   * Left ventricular ejection fraction (LVEF) <50% on screening echocardiogram or multigated acquisition (MUGA) scan.
   * Clinically significant congestive heart failure, unstable angina pectoris,
   * Clinically significant cardiac arrhythmia,
   * Myocardial infarction during the last 6 months, and/or a current electrocardiogram (ECG) tracing that is abnormal in the opinion of the treating Investigator,
   * QTc (QT corrected) prolongation >450 msec (Bazett's Formula), congenitally long QT syndrome, and/or current anti-arrhythmic therapy, has received any marketed or experimental compound in the last 4 weeks prior to entering the study with possible or known effects of QT prolongation, or cumulative high-dose anthracycline therapy.
8. Evidence of clinically significant bradycardia (heart rate <50), or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree AV block (Mobitz Type 2), or patients taking beta blockers, non-dihydropyridine calcium channel blockers, or digoxin.
9. Uncontrolled hypertension (≥140/90 mmHg). Patients who are controlled on antihypertensive medication will be allowed to enter the study.
10. Significant risk for hypokalemia (e.g., patients on high dose diuretics, or with recurrent uncontrolled diarrhea)
11. History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
12. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Current regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
14. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
15. Known to be Human Immunodeficiency Virus (HIV)-positive.
16. Known history of Hepatitis B or C or active Hepatitis A.
17. Symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
18. Treatment with oral corticosteroids (note: inhaled corticosteroids are permitted). IV decadron pre-medication is allowed.
19. Baseline neuropathy of ≥ grade 2.
20. Known allergic reactions to paclitaxel or IV contrast dye despite standard prophylaxis.
21. Patients who require medications that are potent CYP3A4 inhibitors or inducers. Patients who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is longer) prior to the first dose of MK-2206.
22. Patients requiring warfarin therapy. Low molecular weight heparin is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Chien, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled on the study between April 2011 and January 2013. This is a phase one study; the number enrolled was guided by ongoing toxicity assessment.
Pre-assignment Details: 17 patients were initially enrolled; however, one participant experienced rapid progression of disease before receiving any study treatment.
Groups:
- MK-2206: MK-2206 : MK-2206 given orally at a dose of 135 mg weekly Trastuzumab : 2 mg/kg weekly after a 1-time loading dose of 4 mg/kg - trastuzumab Paclitaxel : 80 mg/m2 weekly - paclitaxel
Period: Overall Study
Arm/Group | MK-2206
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all subjects receiving study treatment were included in study analysis
Arm/Group | MK-2206
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 52 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose of MK-2206 Administered Weekly in Combination With Weekly Paclitaxel 80 mg/m^2 and Trastuzumab 2 mg/m^2
Description: The MTD was defined as the dose level resulting in 3 or fewer DLTs in 11 patients, per the modified toxicity probability interval (TPI) method (Ji Y, Li Y, Nebiyou Bekele B: Dose-ﬁnding in phase I clinical trials based on toxicity probability intervals. Clin Trials 4:235-244, 2007), and confirmed in 4 additional patients. Based on interim toxicity data from other studies, the dose was not escalated beyond 135 mg weekly.
Time Frame: 30 days from initiation of dose
Population: Sixteen participants completed at least one cycle of therapy and were evaluable for DLT per protocol. Patients were assessed for DLT during the first 4-week cycle.
Measure: Number; unit: mg
Arm/Group | MK-2206
Number analyzed (Participants) | 16
mg | 135

2. Secondary Outcome: Best Disease Response by Response Evaluation Criteria in Solid Tumor (RECIST), Version 1.1
Description: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufﬁcient shrinkage to qualify for PR nor sufﬁcient increase to qualify for PD, taking as reference the smallest sum diameters while on study
  Non-PR/Non-PD: clinical response of chest wall disease not evaluable by RECIST
Time Frame: 60 days after dose inititation
Population: Analysis included all patients receiving at least 8 weeks of study therapy
Measure: Number; unit: participants
Groups:
- MK-2206: MK-2206 given orally at a dose of 135 mg weekly + Trastuzumab 2 mg/kg weekly after a 1-time loading dose of 4 mg/kg + Paclitaxel 80 mg/m2 weekly
Arm/Group | MK-2206
Number analyzed (Participants) | 16
participants
  Complete Response (CR) | 3
  Partial Response (PR) | 7
  Progressive Disease (PD) | 1
  Stable Disease (SD) | 4
  Non-CR/Non-PD | 1

ADVERSE EVENTS:
Time Frame: 40 weeks
Description: Toxicity assessment continued as long as patient received study treatment; the longest on-study duration was 40 weeks
Arm/Group | MK-2206
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 (N=17)
Liver dysfunction (Hepatobiliary disorders) | 1 (1)
Hemorrhage (General disorders) | 1 (1)
Death (General disorders) | 3 (3) — Death during follow-up (disease progression)
Pain - neuralgia (Nervous system disorders) | 1 (1)
Pain - Abdominal (General disorders) | 1 (2)
Infection with rash grade 3 ANC (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 (N=17)
Anemia (Blood and lymphatic system disorders) | 9 (14) — For all AEs, # participants affected reported here as # events. Patients may have experienced an event more than one time and were clinically managed for recurring toxicity; however, study data are not structured for analysis by patient.
Neutropenia (Blood and lymphatic system disorders) | 14 (30)
Hyperglycemia (Blood and lymphatic system disorders) | 17 (31)
Rash (Skin and subcutaneous tissue disorders) | 15 (24)
Fatigue (General disorders) | 11 (19)
Anorexia/weight loss (General disorders) | 12 (15)
Diarrhea (Gastrointestinal disorders) | 11 (18)
Nausea (General disorders) | 6 (6)
Depression (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Blood and lymphatic system disorders) | 2 (2)
Xerostomia (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent GERD pain (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Hemorrhoid (Gastrointestinal disorders) | 1 (1)
Elevated ALT (Hepatobiliary disorders) | 7 (7)
Elevated AST (Hepatobiliary disorders) | 9 (16)
Hypoalbumenia (Blood and lymphatic system disorders) | 2 (3)
Hyperbilirubin (Hepatobiliary disorders) | 4 (8)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Lower extremity weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Peripheral Neuropathy (Musculoskeletal and connective tissue disorders) | 10 (19)
Stomatitis (Gastrointestinal disorders) | 6 (8)
Altered Taste (General disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Epistaxis (Blood and lymphatic system disorders) | 5 (8)
Hypobilirubin (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 2 (3)
Eye swelling (Eye disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Decreased Hematocrit (Blood and lymphatic system disorders) | 16 (19)
Decreased lymphocytes (Blood and lymphatic system disorders) | 2 (2)
Decreased monocytes (Blood and lymphatic system disorders) | 2 (3)
Decreased RBC (Blood and lymphatic system disorders) | 1 (1)
Decreased WBC (Blood and lymphatic system disorders) | 7 (16)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 8 (15)
Decreased platelets (Blood and lymphatic system disorders) | 4 (7)
Insomnia (General disorders) | 4 (4)
Cracks to fingertips (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (11)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (General disorders) | 2 (2)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Left Calf Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased Potassium (Blood and lymphatic system disorders) | 1 (1)
Decreased Magnesium (Blood and lymphatic system disorders) | 1 (1)
Decreased Calcium (Blood and lymphatic system disorders) | 1 (2)
Elevated BUN (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Groin pain (General disorders) | 1 (1)
Cough (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
MTD was defined as a dose resulting in 3 or fewer DLTs in 11 patients, plus a cohort of 4 patients by a modified TPI dose escalation method. Based on interim toxicity data from other studies, study dose did not exceed 135mg weekly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes